CLINICAL TRIAL: NCT06045429
Title: Effects of Oral Care With 3% Hydrogen Peroxide (Oroxid®) on the Lower Respiratory Tract Microbial Colonisation in Mechanically Ventilated Adult Critically Ill Patients (HyPer-MICROBE Trial); a Single-centre, Randomised, Controlled Trial
Brief Title: Oral Care With 3% Hydrogen Peroxide (Oroxid®) in ICU - Effects on the Lower Airway Microbial Colonisation
Acronym: HyperMICROBE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Jiroutková, Principal Investigator, Kateřina Jiroutková, MD, PhD, EDAIC, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VP/46/0/2022
Record Dates: First submitted 2023-08-24; First posted 2023-09-21 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: VAP - Ventilator Associated Pneumonia
Keywords: pneumonia; hydrogen peroxide; chlorhexidine; respiratory tract microbiome
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia

STUDY DESIGN:
Intervention Model Description: Eligible patients will be recruited in medical-surgical ICU at Kralovske Vinohrady University Hospital (FNKV), managed under an intensivist-led closed ICU, with a 1:1 nurse-to-patient ratio and randomised in equal proportions between 3% hydrogen peroxide arm and 0,2% chlorhexidine digluconate arm.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention nurses can't be blinded to allocation (the mouthwash type - nature of the fluid, its odour etc.), but are strongly inculcated not to disclose the allocation status of the participant at the follow up assessments. As the ICU is paperless and fully computerised, the data in the computer can be acquired and analysed by the researchers without having access to information about the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrogen Peroxide (Experimental): Intervention group: daily oral care will be provided according to the local standard, with 3% hydrogen peroxide, oral assessment and teeth brushing will be completed twice daily (morning and evening).
  Interventions: Drug: Oroxid®
- Chlorhexidine (Active Comparator): Control group: daily oral care will be provided according to the local standard, with 0,2% chlorhexidine, oral assessment and teeth brushing will be completed twice daily (morning and evening).
  Interventions: Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Oroxid® — All patients in experimental arm will receive usual best medical and nursing care with respect to VAP prevention including recently reviewed local "ventilator bundle "; standard microbial surveillance (tracheal aspirate) will be performed twice a week (Monday, Thursday) and always ad hoc according to the clinical situation. This reflects current practice. Daily oral care will be provided using Oroxid® mouthwash.
  Other Names: 3% hydrogen peroxide mouthwash
  Arms: Hydrogen Peroxide
Drug: Chlorhexidine mouthwash — All patients in experimental arm will receive usual best medical and nursing care with respect to VAP prevention including recently reviewed local "ventilator bundle "; standard microbial surveillance (tracheal aspirate) will be performed twice a week (Monday, Thursday) and always ad hoc according to the clinical situation. This reflects current practice. Daily oral care will be provided using 0,2% chlorhexidine
  Other Names: 0,2% chlorhexidine gluconate
  Arms: Chlorhexidine

SUMMARY:
HyPerMICROBE is a single-centre, controlled, randomised, prospective, superiority clinical trial to compare the efficacy of daily oral care with 3% hydrogen peroxide (Oroxid®) versus standard of care (0.2% chlorhexidine digluconate) on the cumulative incidence of lower respiratory tract microbial colonisation in mechanically ventilated adult critically ill patients.

DETAILED DESCRIPTION:
Rationale: Ventilator-associated pneumonia (VAP) is the most common hospital-acquired infection (HAI) in the intensive care unit (ICU), and its impact is very high in terms of morbidity, length of hospital stay and overall costs. Chlorhexidine for oral care in critically ill has no clear impact on VAP rates and may cause harm. 3% hydrogen peroxide (Oroxid) could be a promising substitute.

Aim: To test effectivity and safety of 3% hydrogen peroxide solution on ventilator-associated complications

Design: Prospective, single center, parallel group randomised controlled trial. Subjects: ICU patients (general ICU)

Treatment in the intervention group: daily oral care with 3% hydrogen peroxide

Control group: Standard-of-care protocolised daily oral care with 0,2% chlorhexidine

Primary outcome: Cumulative incidence of lower respiratory tract microbial colonisation analysed by Kaplan-Maier method, censored in the case of ICU discharge or extubation > 24h.

Secondary and exploratory outcomes: Differences in the relative risk of infection related ventilator-associated complications, antibiotic (ATB) consumption analysis, intraoral complications, reported using the Bedside oral exam (BOE) score, validated and adopted for ICU, length of ICU stay in days (time frame: at 3 months), number of ventilator-free days (time frame: at 28 days); that is, number of days, out of 28 days after admission, that patient has not been supported by mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. In-patient of ICU and expected to stay > 5 days
3. Mechanical ventilation or imminent need of it; predicted length of mechanical ventilation (MV) ≥ 72h
4. Clinical Pulmonary Infection score (CPIS) less than 6 at the baseline
5. No history and symptoms of aspiration at the baseline

Exclusion Criteria:

1. ATB therapy of respiratory infection on admission
2. Suspected pulmonary infection on admission and in the first 48h of mechanical ventilation
3. Pregnancy
4. Oral ulcers or injuries
5. Patient with a history of hydrogen peroxide allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of lower respiratory tract microbial colonisation analysed by Kaplan-Maier method, censored in the case of ICU discharge or extubation > 24h. | 18 months
  To detect microorganisms in the lower respiratory tract, tracheal aspirate will be directly cultured for detecting Gram-positive, Gram-negative, and anaerobic bacteria and fungi. Standard microbial surveillance (tracheal aspirate) will be performed on admission, twice a week (Monday, Thursday) and always ad hoc according to the clinical situation.

SECONDARY OUTCOMES:
Differences in the relative risk of infection related ventilator associated complications (IVAC) | 18 months
  According to the Centers for Disease Control and Prevention (CDC) criteria, the IVAC diagnosis will be established based on:
  * an increase of the daily minimum positive end-expiratory pressure (PEEP) of ≥3 cm H2O and/or the daily minimum inspired oxygen fraction (FiO2) of ≥20 points sustained for ≥2 days and
  * an evidence of a new infection present (abnormal temperature or white blood cell count) and prescription of a new antibiotic for ≥4 days
ATB exposure at discharge | From the date of enrolment through to the date of ICU discharge, approximately 28 days
  Duration of antibiotics prescribed at discharge
Intraoral complications, reported using the Bedside oral exam (BOE) score, validated and adopted for ICU. | will be measured at 24 hours (T1), day 3 (T2), day 7 (T3) and day 14 (T4) after admission
  BOE score ranges from 8 (excellent oral health) to 24 (poor oral health). The BOE scores ranging from 8-10 are considered as indicative of excellent oral health, from 11-14 as moderately impaired oral health and from 15-24 as significantly impaired oral health
Length of ICU stay in days | at 3 months
  that is, length of ICU stay in days
Number of ventilator-free days; | at 28 days
  that is, number of days, out of 28 days after admission, that patient has not been supported by mechanical ventilation

OTHER OUTCOMES:
Composition of the oral and lower airway microbiome between groups measured by the bacterial 16S rRNA sequencing | day 0, day 7 and day 14
  Microbial DNA will be sequentially (on admission, day 3, 7 and 14) sampled and isolated from prespecified sites in oral cavity, hypopharynx and lower respiratory tract. Microbial DNA will be analyzed by 16S rRNA amplicon sequencing and quantified by multiplex qPCR method. Paired comparison of bacteriomes between intervention group and control group will be performed to identify potentially risky host bacteriome profiles.
Antibiotic Free Days | up to 30 days
  The number of days where participant did not require the use of antibiotics
The number of participants with Non-pulmonary infections | up to 30 days
  The number of participants with Non-pulmonary infections

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Jiroutková, MD, Principal Investigator — 3rd Faculty of Medicine, Charles University and FNKV, Prague
Locations (1):
- 3rd Faculty of Medicine and FNKV, Prague, Czechia